CLINICAL TRIAL: NCT06767436
Title: A Multi-center Cohort Study to Evaluate the Real-world Efficacy and Safety of Trastuzumab-deruxtecan in Advanced Gastric Cancer
Brief Title: A Multi-center Real-world Efficacy and Safety of Trastuzumab-deruxtecan in Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Minkyu Jung, Principal Investigator, Yonsei University
Other Study IDs: 4-2024-1144
Record Dates: First submitted 2024-12-26; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Trastuzumab-deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Institutions will be selected
* This study aims to collect real-world data, targeting patients who started treatment with Enhertu from September 2022, for clinical data collection
* Among patients treated with Enhertu, those who have passed away or are no longer visiting due to hospice care will have their clinical data collected without consent until August 19, 2024
* For patients who are scheduled to receive Enhertu treatment, are currently undergoing treatment, or have previously undergone treatment but experienced disease progression and are now receiving subsequent chemotherapy (i.e., patients with newly added data after registration)
* Efficacy evaluation

DETAILED DESCRIPTION:
* Institutions will be selected through the Gastric Cancer Subcommittee of the Korean Cancer Study Group.
* This study aims to collect real-world data, targeting patients who started treatment with trastuzumab-deruxtecan from September 2022, for clinical data collection.
* Among patients treated with trastuzumab-deruxtecan, those who have passed away or are no longer visiting due to hospice care will have their clinical data collected without consent until August 19, 2024.
* For patients who are scheduled to receive Enhertu treatment, are currently undergoing treatment, or have previously undergone treatment but experienced disease progression and are now receiving subsequent chemotherapy (i.e., patients with newly added data after registration), data will be collected with consent until March 31, 2027.
* Efficacy evaluation will include overall survival (OS), progression-free survival (PFS), and tumor response rate (TRR)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older.
* Patients with pathologically confirmed metastatic, recurrent, or unresectable gastric/gastroesophageal adenocarcinoma.
* Patients whose tumor tissue shows HER2 immunohistochemistry (IHC) results of 3+ or 2+ with in-situ hybridization (ISH) positivity.
* Patients who received Trastuzumab Deruxtecan as third-line or later treatment.

Exclusion Criteria:

* Patients with HER2-negative gastric cancer.
* Patients who did not provide consent to participate in the study.
* Patients who received Trastuzumab Deruxtecan as first-line or second-line treatment as part of a clinical trial.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Institutions will be selected
  * targeting patients who started treatment with Enhertu from September 2022, for clinical data collection
  * Among patients treated with Enhertu, those who have passed away or are no longer visiting due to hospice care will have their clinical data collected without consent until August 19, 2024.
  * For patients who are scheduled to receive Enhertu treatment, are currently undergoing treatment, or have previously undergone treatment but experienced disease progression and are now receiving subsequent chemotherapy (i.e., patients with newly added data after registration), data will be collected with consent until March 31, 2027.
  * Efficacy evaluation will include overall survival (OS), progression-free survival (PFS), and tumor response rate (TRR)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11-04 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 1 year
  To present real-world clinical outcomes of trastuzumab-deruxtecan as third-line or later treatment in HER2-positive gastric cancer.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE V5.0
analyze the correlation | 1 year
  To analyze the correlation between HER2 immunohistochemistry (IHC) results and the efficacy of trastuzumab-deruxtecan.

CONTACTS AND LOCATIONS:
Overall Officials: minkyu Jung, Principal Investigator — Yonsei Cencer center
Locations (1):
- minkyu Jung, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Shitara K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Yamaguchi K; DESTINY-Gastric01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Gastric Cancer. N Engl J Med. 2020 Jun 18;382(25):2419-2430. doi: 10.1056/NEJMoa2004413. Epub 2020 May 29. PMID 32469182